CLINICAL TRIAL: NCT00345176
Title: Age-Related Eye Disease Study 2 (AREDS2): A Multi-center, Randomized Trial of Lutein, Zeaxanthin and Omega-3 Long-Chain Polyunsaturated Fatty Acids (Docosahexaenoic Acid [DHA] and Eicosapentaenoic Acid [EPA]) in Age-Related Macular Degeneration
Brief Title: Age-Related Eye Disease Study 2 (AREDS2)
Acronym: AREDS2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Office of Dietary Supplements (ODS) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEI-120; N01-EY-5-0007 (Other Grant/Funding Number: NIH); HHS-N-260-2005-00007-C (Other Grant/Funding Number: HHS); CC-070025 (Other: NIH Clinical Center); 07-EI-0025 (Other: National Eye Institute); NCT00409513 (obsolete NCT alias)
Record Dates: First submitted 2006-06-14; First posted 2006-06-27 (Estimated); Results first posted 2013-12-24 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-04

CONDITIONS: Age-related Macular Degeneration; Cataract
Keywords: age-related macular degeneration; AMD; lutein; zeaxanthin; docosahexaenoic acid; eicosapentaenoic acid
MeSH Terms: conditions — Macular Degeneration; Cataract | interventions — Lutein; Zeaxanthins; Docosahexaenoic Acids; Eicosapentaenoic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lutein/Zeaxanthin (Active Comparator): lutein (10mg)/zeaxanthin (2 mg)
  Interventions: Dietary Supplement: Lutein/zeaxanthin
- DHA/EPA (Active Comparator): DHA (350 mg)/EPA (650 mg)
  Interventions: Dietary Supplement: DHA/EPA
- Lutein/Zeaxanthin + DHA/EPA (Active Comparator): lutein (10 mg)/zeaxanthin (2 mg) + DHA (350 mg)/EPA (650 mg)
  Interventions: Drug: Lutein/zeaxanthin and DHA/EPA
- Placebo/Control (Placebo Comparator): Considered control because all participants received the AREDS formulation

INTERVENTIONS:
Dietary Supplement: Lutein/zeaxanthin — 10 mg lutein and 2 mg zeaxanthin (1 tablet) Placebo-DHA/EPA (2 soft-gel capsules)
  Arms: Lutein/Zeaxanthin
Dietary Supplement: DHA/EPA — Placebo-lutein/zeaxanthin (1 tablet) 350 mg DHA and 650 mg EPA (2 soft-gel capsules)
  Other Names: docosahexaenoic acid; eicosapentaenoic acid
  Arms: DHA/EPA
Drug: Lutein/zeaxanthin and DHA/EPA — 10 mg lutein and 2 mg zeaxanthin (1 tablet) 350 mg DHA and 650 mg EPA (2 soft-gel capsules)
  Arms: Lutein/Zeaxanthin + DHA/EPA

SUMMARY:
Oral supplementation with the Age-Related Eye Disease Study (AREDS) formulation (antioxidant vitamins C and E, beta carotene, and zinc) has been shown to reduce the risk of progression to advanced age-related macular degeneration (AMD). Observational data suggest that increased dietary intake of lutein + zeaxanthin (carotenoids), omega-3 long-chain polyunsaturated fatty acids (docosahexaenoic acid [DHA] + eicosapentaenoic acid [EPA]), or both might further reduce this risk. AREDS2 was designed to test whether adding lutein + zeaxanthin, DHA + EPA, or lutein + zeaxanthin and DHA + EPA to the AREDS formulation might further reduce the risk of progression to advanced AMD. A secondary goal was to test the effects of eliminating beta carotene and reducing zinc dose in the AREDS formulation.

DETAILED DESCRIPTION:
AREDS2 was a randomized, double-masked, placebo-controlled, 2x2 factorial trial evaluating the risks and benefits of adding lutein (10 mg) + zeaxanthin (2 mg), DHA (350 mg) + EPA (650 mg), or both to the AREDS formulation, which consisted of vitamins C (500 mg), vitamin E (400 international units), beta carotene (15 mg), zinc (80 mg as zinc oxide), and copper (2 mg as cupric oxide) for the treatment of progression to advanced AMD. The study enrolled 4,203 participants aged 50 to 85 years, with sufficiently clear ocular media to allow accurate assessment of AMD from fundus photographs. Subjects were enrolled on the basis of the AREDS Simplified Severity Scale for defining risk categories for development of advanced age-related macular degeneration. All participants were offered additional treatment with the original AREDS formulation (now considered standard of care) and 3 variations of this formula. These are: (1) no beta-carotene; (2) lower amount of zinc (25 mg); and (3) no beta-carotene and lower amount of zinc (25 mg). Eligible participants were followed for a minimum of five years.

Multiple ancillary studies were conducted using the parent study (AREDS2) data to explore:

1. Effects of oral supplementation of omega-3 fatty acids, lutein/zeaxanthin, zinc, and beta-carotene on cognitive function

   1. Outcome is measured with a battery of tests administered over the telephone at baseline, and at years 2 and 4 of the study.
   2. Primary outcome is the change in the composite score for the results of the cognitive function testing from baseline over time.
2. Effects of oral supplementation of omega-3 fatty acids, lutein/zeaxanthin on cardiovascular disease

   a. Primary measure of cardiovascular morbidity and mortality
3. Effects of oral supplementation of omega-3 fatty acids, lutein/zeaxanthin on the peripheral retina

   a. Primary outcome is the development of peripheral drusen, geographic atrophy, reticular pigmentary changes, and pseudoreticular drusen.
4. Association of genotype polymorphisms with age-related macular degeneration and cataract

   a. Whole genome sequencing will be completed. Evaluation of association genetic associations with disease will be conducted using AREDS controls.
5. Association of genotype polymorphisms with progression of age-related macular degeneration

   a. Whole genome sequencing is conducted. Progression from early to late and severe stages of AMD will be examined with the genotype data to evaluate the risks of progression associated with the genotype polymorphisms.
6. Association of genotype polymorphisms with dietary intake a. Whole genome sequencing is conducted. Progression from early to late and severe stages of AMD will be examined regarding potential interaction of the dietary intake with the genotype data to evaluate the risks of progression.
7. Association of genotype polymorphisms with AREDS2 supplements a. Interaction of genetic polymorphisms with AREDS2 supplements for progression to late AMD will be evaluated using the data from the whole genome sequencing project.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 50 and 85 years
* Macular status ranges from large drusen in both eyes or large drusen in one eye and advanced AMD (neovascular AMD or geographic atrophy) in the fellow eye

Exclusion Criteria:

* Ocular media not clear enough to allow good fundus photography

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4203 (Actual)
Dates: Start 2006-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Y Chew, MD, Study Chair — National Eye Institute, National Institutes of Health; John Paul SanGiovanni, Sc.D., Study Director — National Eye Institute, National Institutes of Health
Locations (91):
- United States (91):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Jones Eye Institute - UAMS, Little Rock, Arkansas
  - Retina-Vitreous Associates Medical Group, Beverly Hills, California
  - Shiley Eye Center - UCSD, La Jolla, California
  - Loma Linda University, Loma Linda, California
  - Doheny Eye Institute, Los Angeles, California
  - Jules Stein Eye Institute, Los Angeles, California
  - VA Northern California Health Care System, Martinez, California
  - Southern California Desert Retina Consultants, MC, Palm Springs, California
  - University of California, Davis, Sacramento, California
  - West Coast Retina Medical Group, Inc, San Francisco, California
  - Pacific Eye Associates, San Francisco, California
  - Colorado Retina Associates, Denver, Colorado
  - Eldorado Retina Associates, PC, Louisville, Colorado
  - Yale University Eye Center, New Haven, Connecticut
  - Retina Group of Florida, Fort Lauderdale, Florida
  - University of Florida, Jacksonville, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Emory University Eye Center, Atlanta, Georgia
  - Georgia Retina, PC, Decatur, Georgia
  - Northwestern University, Chicago, Illinois
  - The University of Illinois, Chicago, Illinois
  - NorthShore University HealthSystems, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - University of Iowa, Iowa City, Iowa
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Paducah Retinal Center, Paducah, Kentucky
  - Elman Retina Group, Baltimore, Maryland
  - Wilmer Eye Institute, Johns Hopkins Hospital, Baltimore, Maryland
  - National Eye Institute, Bethesda, Maryland
  - The Retina Group of Washington, Chevy Chase, Maryland
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Kresge Eye Institute, Detroit, Michigan
  - Henry Ford Health System - Eye Care Services, Detroit, Michigan
  - Vision Research Foundation, Grand Rapids, Michigan
  - Vision Research Foundation, Royal Oak, Michigan
  - Vision Research Foundation, Traverse City, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University Health Care - Mason Eye Institute, Columbia, Missouri
  - Eye Foundation of Kansas City, Kansas City, Missouri
  - Mid-America Retina Consultants, PA, Kansas City, Missouri
  - The Retina Institute, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Delaware Valley Retina Associates, Lawrenceville, New Jersey
  - UMDNJ, Newark, New Jersey
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - New York Eye and Ear Infirmary, New York, New York
  - Manhattan Eye, Ear and Throat Hospital, New York, New York
  - University of Rochester Eye Institute, Rochester, New York
  - Retina Consultants, PLLC, Slingerlands, New York
  - The Research Foundation of SUNY/Stony Brook, Stony Brook, New York
  - Western Carolina Retinal Associates, Asheville, North Carolina
  - UNC Department of Ophthalmology, Chapel Hill, North Carolina
  - Charlotte Eye Ear Nose and Throat Associates, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Wake Forest University Eye Center, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Retina Associates of Cleveland, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Retina Associates of Cleveland, Middleburg Heights, Ohio
  - Retina Associates of Cleveland, Youngstown, Ohio
  - Dean McGee Eye Institute, Oklahoma City, Oklahoma
  - Devers Eye Institute, Portland, Oregon
  - Retina Northwest, PC, Portland, Oregon
  - Pennsylvania Retina Specialists, PC, Camp Hill, Pennsylvania
  - Penn State M.S. Hershey Medical Center, Hershey, Pennsylvania
  - Scheie Eye Institute, Philadelphia, Pennsylvania
  - Wills Eye Hospital/Mid Atlantic Retina, Philadelphia, Pennsylvania
  - Retina Vitreous Consultants, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Palmetto Retina Center, Columbia, South Carolina
  - Carolina Retina Center, Columbia, South Carolina
  - Southeastern Retina Associates, PC, Knoxville, Tennessee
  - University of Tennessee, Memphis, Tennessee
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - Texas Retina Associates, Arlington, Texas
  - Texas Retina Associates, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Retina Consultants of Houston, Houston, Texas
  - Texas Retina Associates, Lubbock, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - John Moran Eye Center, Salt Lake City, Utah
  - Fletcher Allen Health Care, Burlington, Vermont
  - The Retina Group of Washington, Fairfax, Virginia
  - Retina Center Northwest, Silverdale, Washington
  - University of Wisconsin, Madison, Wisconsin
  - The Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Evans JR, Lawrenson JG. Antioxidant vitamin and mineral supplements for slowing the progression of age-related macular degeneration. Cochrane Database Syst Rev. 2023 Sep 13;9(9):CD000254. doi: 10.1002/14651858.CD000254.pub5. PMID 37702300
- [Derived] Bhandari S, Vitale S, Agron E, Clemons TE, Chew EY; Age-Related Eye Disease Study 2 Research Group. Cataract Surgery and the Risk of Developing Late Age-Related Macular Degeneration: The Age-Related Eye Disease Study 2 Report Number 27. Ophthalmology. 2022 Apr;129(4):414-420. doi: 10.1016/j.ophtha.2021.11.014. Epub 2021 Nov 16. PMID 34793832
- [Derived] Keenan TD, Agron E, Mares JA, Clemons TE, van Asten F, Swaroop A, Chew EY; AREDS and AREDS2 Research Groups. Adherence to a Mediterranean diet and cognitive function in the Age-Related Eye Disease Studies 1 & 2. Alzheimers Dement. 2020 Jun;16(6):831-842. doi: 10.1002/alz.12077. Epub 2020 Apr 13. PMID 32285590
- [Derived] Chew EY, Clemons TE, Agron E, Launer LJ, Grodstein F, Bernstein PS; Age-Related Eye Disease Study 2 (AREDS2) Research Group. Effect of Omega-3 Fatty Acids, Lutein/Zeaxanthin, or Other Nutrient Supplementation on Cognitive Function: The AREDS2 Randomized Clinical Trial. JAMA. 2015 Aug 25;314(8):791-801. doi: 10.1001/jama.2015.9677. PMID 26305649
- [Derived] Writing Group for the AREDS2 Research Group; Bonds DE, Harrington M, Worrall BB, Bertoni AG, Eaton CB, Hsia J, Robinson J, Clemons TE, Fine LJ, Chew EY. Effect of long-chain omega-3 fatty acids and lutein + zeaxanthin supplements on cardiovascular outcomes: results of the Age-Related Eye Disease Study 2 (AREDS2) randomized clinical trial. JAMA Intern Med. 2014 May;174(5):763-71. doi: 10.1001/jamainternmed.2014.328. PMID 24638908
- [Derived] Age-Related Eye Disease Study 2 (AREDS2) Research Group; Chew EY, Clemons TE, Sangiovanni JP, Danis RP, Ferris FL 3rd, Elman MJ, Antoszyk AN, Ruby AJ, Orth D, Bressler SB, Fish GE, Hubbard GB, Klein ML, Chandra SR, Blodi BA, Domalpally A, Friberg T, Wong WT, Rosenfeld PJ, Agron E, Toth CA, Bernstein PS, Sperduto RD. Secondary analyses of the effects of lutein/zeaxanthin on age-related macular degeneration progression: AREDS2 report No. 3. JAMA Ophthalmol. 2014 Feb;132(2):142-9. doi: 10.1001/jamaophthalmol.2013.7376. PMID 24310343
- [Derived] Domalpally A, Danis RP, Chew EY, Clemons TE, Reed S, Sangiovanni JP, Ferris FL 3rd; Age-Related Eye Disease Study 2 Research Group. Evaluation of optimized digital fundus reflex photographs for lens opacities in the age-related eye disease study 2: AREDS2 report 7. Invest Ophthalmol Vis Sci. 2013 Sep 5;54(9):5989-94. doi: 10.1167/iovs.13-12301. PMID 23887802
- [Derived] Toy BC, Krishnadev N, Indaram M, Cunningham D, Cukras CA, Chew EY, Wong WT. Drusen regression is associated with local changes in fundus autofluorescence in intermediate age-related macular degeneration. Am J Ophthalmol. 2013 Sep;156(3):532-542.e1. doi: 10.1016/j.ajo.2013.04.031. Epub 2013 Jul 3. PMID 23830564
- [Derived] Age-Related Eye Disease Study 2 (AREDS2) Research Group; Chew EY, SanGiovanni JP, Ferris FL, Wong WT, Agron E, Clemons TE, Sperduto R, Danis R, Chandra SR, Blodi BA, Domalpally A, Elman MJ, Antoszyk AN, Ruby AJ, Orth D, Bressler SB, Fish GE, Hubbard GB, Klein ML, Friberg TR, Rosenfeld PJ, Toth CA, Bernstein P. Lutein/zeaxanthin for the treatment of age-related cataract: AREDS2 randomized trial report no. 4. JAMA Ophthalmol. 2013 Jul;131(7):843-50. doi: 10.1001/jamaophthalmol.2013.4412. PMID 23645227
- [Derived] Age-Related Eye Disease Study 2 Research Group. Lutein + zeaxanthin and omega-3 fatty acids for age-related macular degeneration: the Age-Related Eye Disease Study 2 (AREDS2) randomized clinical trial. JAMA. 2013 May 15;309(19):2005-15. doi: 10.1001/jama.2013.4997. PMID 23644932
- [Derived] Danis RP, Domalpally A, Chew EY, Clemons TE, Armstrong J, SanGiovanni JP, Ferris FL 3rd; AREDS2 Study Group. Methods and reproducibility of grading optimized digital color fundus photographs in the Age-Related Eye Disease Study 2 (AREDS2 Report Number 2). Invest Ophthalmol Vis Sci. 2013 Jul 8;54(7):4548-54. doi: 10.1167/iovs.13-11804. PMID 23620429
- [Derived] Bernstein PS, Ahmed F, Liu A, Allman S, Sheng X, Sharifzadeh M, Ermakov I, Gellermann W. Macular pigment imaging in AREDS2 participants: an ancillary study of AREDS2 subjects enrolled at the Moran Eye Center. Invest Ophthalmol Vis Sci. 2012 Sep 14;53(10):6178-86. doi: 10.1167/iovs.12-10275. PMID 22879423
- [Derived] Hubbard LD, Danis RP, Neider MW, Thayer DW, Wabers HD, White JK, Pugliese AJ, Pugliese MF; Age-Related Eye Disease 2 Research Group. Brightness, contrast, and color balance of digital versus film retinal images in the age-related eye disease study 2. Invest Ophthalmol Vis Sci. 2008 Aug;49(8):3269-82. doi: 10.1167/iovs.07-1267. Epub 2008 Apr 17. PMID 18421079
- See also: NEI Website: Age-Related Eye Disease Study 2 — http://www.nei.nih.gov/areds2/
- See also: AREDS2 Website — http://www.areds2.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 2006 and September 2008 a total of 4,203 participants aged 50 - 85 years were randomized at 82 clinical sites.
Pre-assignment Details: Prior to randomization, participants had to complete the Qualification phase. They could only be randomized if they took at least 75% of the run-in medication.
Period: Overall Study
Arm/Group | Placebo/Control | Lutein/Zeaxanthin | DHA/EPA | Lutein/Zeaxanthin + DHA/EPA
Started | 1012 | 1044 | 1068 | 1079
Completed | 1007 | 1038 | 1062 | 1069
Not Completed | 5 | 6 | 6 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Control | Lutein/Zeaxanthin | DHA/EPA | Lutein/Zeaxanthin + DHA/EPA | Total
Number analyzed (Participants) | 1012 | 1044 | 1068 | 1079 | 4203
Age, Continuous [Median (Inter-Quartile Range); unit: Participants] | 74 [68 to 79] | 74 [68 to 79] | 74 [68 to 79] | 75 [68 to 79] | 74 [68 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 548 | 596 | 603 | 641 | 2388
  Male | 464 | 448 | 465 | 438 | 1815

OUTCOME MEASURES:

1. Primary Outcome: Development of Advanced AMD in People at Moderate to High Risk for Progression.
Description: Defined as central geographic atrophy or retinal features of choroidal neovascularization detected on central grading of the stereoscopic fundus photographs or a history of treatment for advanced AMD after study enrollment.
Time Frame: 5 years of follow-up
Population: Intention to Treat. Participants lost to follow-up during the course of the study were censored at the time of last contact.
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Placebo/Control | Lutein/Zeaxanthin | DHA/EPA | Lutein/Zeaxanthin + DHA/EPA
Number analyzed (Participants) | 1007 | 1038 | 1062 | 1069
Number analyzed (Eyes) | 1691 | 1709 | 1749 | 1742
Eyes | 493 | 468 | 507 | 472
Statistical Analysis 1: Comparison: Placebo/Control vs Lutein/Zeaxanthin; Each of the 3 active arms was compared to the placebo/control arm; Test type: Superiority or Other; p < 0.013, Regression, Cox — Adjusted for 3 treatment versus placebo comparisons and interim analyses; Adjusted for baseline AMD status; Hazard Ratio (HR) = 0.90, 98.7% CI 2-sided [0.76 to 1.07] — The reference group is placebo
Statistical Analysis 2: Comparison: Placebo/Control vs DHA/EPA; Test type: Superiority or Other; p < 0.013, Regression, Cox — Adjusted for multiple comparisons; Hazard Ratio (HR) = 0.97, 98.7% CI 2-sided [0.82 to 1.16]
Statistical Analysis 3: Comparison: Placebo/Control vs Lutein/Zeaxanthin + DHA/EPA; Test type: Superiority or Other; p < 0.013, Regression, Cox; Adjusted for multiple comparisons; Hazard Ratio (HR) = 0.89, 98.7% CI 2-sided [0.75 to 1.06]

2. Secondary Outcome: Progression to Moderate Vision Loss
Description: Loss defined as >/= 3 lines of letters from baseline or treatment for choroidal neovascularization
Time Frame: 5 years of follow-up
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Placebo/Control | Lutein/Zeaxanthin | DHA/EPA | Lutein/Zeaxanthin + DHA/EPA
Number analyzed (Participants) | 1007 | 1038 | 1062 | 1069
Number analyzed (Eyes) | 1630 | 1660 | 1694 | 1672
Eyes | 515 | 509 | 519 | 506
Statistical Analysis 1: Comparison: Placebo/Control vs Lutein/Zeaxanthin; Test type: Superiority or Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.84 to 1.08]
Statistical Analysis 2: Comparison: Placebo/Control vs DHA/EPA; Test type: Superiority or Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.84 to 1.09]
Statistical Analysis 3: Comparison: Placebo/Control vs Lutein/Zeaxanthin + DHA/EPA; Test type: Superiority or Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.83 to 1.07]

3. Secondary Outcome: Adverse Events
Description: Safety outcomes included serious adverse events and mortality.
Time Frame: 5 years of follow-up
Population: Number of deaths in 5 years
Measure: Number; unit: Participants
Arm/Group | Placebo/Control | Lutein/Zeaxanthin | DHA/EPA | Lutein/Zeaxanthin + DHA/EPA
Number analyzed (Participants) | 1012 | 1044 | 1068 | 1079
Participants
  Mortality | 81 | 87 | 96 | 104
  Serious Adverse Events | 479 | 484 | 505 | 519
Statistical Analysis 1: Comparison: Placebo/Control vs Lutein/Zeaxanthin; Comparison of Lutein/Zeaxantin versus Control for mortality; Test type: Superiority or Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.77 to 1.40]
Statistical Analysis 2: Comparison: Placebo/Control vs DHA/EPA; Comparison of DHA/EPA versus Placebo for mortality; Test type: Superiority or Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.84 to 1.52]
Statistical Analysis 3: Comparison: Placebo/Control vs Lutein/Zeaxanthin + DHA/EPA; Comparison of Lutein/Zeaxanthin + DHA/EPA versus Placebo for Mortality; Test type: Superiority or Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.92 to 1.65]

4. Secondary Outcome: Progression to Cataract Surgery
Description: The study examined the effects of lutein/zeaxanthin on progression to cataract surgery with data collected during regular telephone contacts and the annual study visits.
Time Frame: 5 years of follow-up
Population: Includes participants who were phakic in at least 1 eye at baseline
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Groups:
- No Lutein/Zeaxanthin: Lutein main effect - includes participants who did not receive Lutein/Zeaxanthin
- Lutein/Zeaxanthin: Lutein main effect - includes all participants who received Lutein/Zeaxanthin
Arm/Group | No Lutein/Zeaxanthin | Lutein/Zeaxanthin
Number analyzed (Participants) | 1577 | 1578
Number analyzed (Eyes) | 3022 | 3005
Eyes | 708 | 681
Statistical Analysis 1: Comparison: No Lutein/Zeaxanthin vs Lutein/Zeaxanthin; Test type: Superiority or Other; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.84 to 1.10]

5. Other Pre Specified Outcome: Incident Cardiovascular Disease
Description: Effects of oral supplementation of omega-3 fatty acids, lutein/zeaxanthin on cardiovascular disease
Time Frame: 5 years of follow-up
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Cognition as Measured by a Telephone Battery
Description: Effects of oral supplementation of omega-3 fatty acids, lutein/zeaxanthin, zinc, and beta-carotene on cognitive function
Time Frame: 5 years of follow-up
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Prevalence of Peripheral Changes as Measured Using OPTOS Imaging
Description: Effects of oral supplementation of omega-3 fatty acids, lutein/zeaxanthin on the peripheral retina
Time Frame: 5 years of follow-up
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Genetics for the Association of AMD and Cataract
Time Frame: 5 years of follow-up
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Genetics for the Progression of AMD and Cataract
Time Frame: 5 years of follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 years
Description: Adverse events reported by System Organ Class
Arm/Group | Placebo/Control | Lutein/Zeaxanthin | DHA/EPA | Lutein/Zeaxanthin + DHA/EPA
Serious Adverse Events (participants affected / at risk) | 479/1012 | 484/1044 | 505/1068 | 519/1079
Other Adverse Events (participants affected / at risk) | 717/1012 | 791/1044 | 759/1068 | 791/1079
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Control (N=1012) | Lutein/Zeaxanthin (N=1044) | DHA/EPA (N=1068) | Lutein/Zeaxanthin + DHA/EPA (N=1079)
Cardiac Disorders (Cardiac disorders) | 96 (122) | 110 (138) | 119 (144) | 103 (133)
Gastrointestinal disorders (Gastrointestinal disorders) | 76 (101) | 69 (81) | 58 (72) | 61 (71)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 12 (14) | 11 (11) | 9 (10) | 7 (7)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 7 (7) | 3 (3) | 4 (4) | 1 (1)
Congenital, familian and genetic disorders (Congenital, familial and genetic disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Endocrine disorders (Endocrine disorders) | 2 (2) | 3 (3) | 3 (3) | 0 (0)
Eye disorders (Eye disorders) | 3 (3) | 11 (13) | 4 (6) | 0 (0)
General disorders and administration site conditions (General disorders) | 54 (60) | 50 (54) | 51 (58) | 46 (50)
Hepatobiliary disorders (Hepatobiliary disorders) | 8 (8) | 16 (16) | 16 (16) | 17 (18)
Immune system disorders (Immune system disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Infections and infestations (Infections and infestations) | 90 (109) | 102 (139) | 103 (144) | 99 (127)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 76 (90) | 62 (72) | 74 (90) | 66 (84)
Investigations (Investigations) | 14 (14) | 19 (20) | 13 (15) | 12 (12)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 21 (22) | 16 (18) | 13 (13) | 23 (25)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 66 (77) | 74 (91) | 71 (85) | 85 (101)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 80 (103) | 88 (111) | 83 (100) | 92 (112)
Nervous system disorders (Nervous system disorders) | 66 (73) | 74 (93) | 72 (87) | 73 (86)
Psychiatric disorders (Psychiatric disorders) | 4 (4) | 5 (5) | 5 (5) | 9 (11)
Renal and urinary disorders (Renal and urinary disorders) | 19 (20) | 25 (26) | 24 (25) | 25 (29)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 9 (11) | 8 (8) | 12 (13) | 11 (11)
Respioratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 44 (59) | 43 (52) | 37 (50) | 46 (51)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (7) | 3 (3) | 5 (5)
Surgical and medical procedures (Surgical and medical procedures) | 32 (32) | 29 (31) | 27 (30) | 32 (32)
Vascular disorders (Vascular disorders) | 41 (45) | 40 (42) | 42 (45) | 42 (46)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/Control (N=1012) | Lutein/Zeaxanthin (N=1044) | DHA/EPA (N=1068) | Lutein/Zeaxanthin + DHA/EPA (N=1079)
Dry eye (Eye disorders) | 55 (62) | 39 (40) | 64 (70) | 62 (70)
Eye disorder (Eye disorders) | 67 (100) | 67 (96) | 62 (98) | 82 (152)
Visual disturbance (Eye disorders) | 88 (118) | 110 (139) | 84 (116) | 88 (119)
Vitreous disorder (Eye disorders) | 133 (208) | 154 (213) | 165 (228) | 162 (208)
Change in bowel habit (Gastrointestinal disorders) | 57 (69) | 67 (77) | 48 (58) | 57 (60)
Bronchitis (Infections and infestations) | 62 (72) | 69 (83) | 57 (80) | 56 (66)
Upper respiratory tract infection (Infections and infestations) | 139 (175) | 150 (190) | 139 (179) | 138 (173)
Urinary tract infection (Infections and infestations) | 57 (82) | 75 (103) | 71 (108) | 73 (96)
Hypertension (Vascular disorders) | 59 (66) | 60 (62) | 69 (72) | 73 (73)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No